CLINICAL TRIAL: NCT03667183
Title: Levels of Body Composition, Energy Expenditure, Physical Fitness and Quality of Life in Adolescents With Eating Disorders: Effect of a Pilates Program
Brief Title: Pilates Program in Female Adolescent With Eating Disorders
Acronym: PITCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pablo de Olavide (Other)
Collaborators: Complejo Hospitalario Universitario de Huelva (Other)
Responsible Party: Principal Investigator, Sofía Mª Martínez Sánchez, Principal Investigator, Universidad Pablo de Olavide
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UniversidadPO
Record Dates: First submitted 2018-09-05; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Eating Disorder; Female Adolescents
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilates Group (Experimental): Female adolescents with eating disorders who receive Pilates for 10 weeks.
  Interventions: Other: Pilates

INTERVENTIONS:
Other: Pilates — Specific postures in movement according to Pilates guidelines.

SUMMARY:
Physical exercise helps patients with eating disorders by improving their physical fitness, quality of life and other specific variables of this pathology. Pilates has a beneficial effect both physically and mentally on healthy population and other diseases. In patients with eating disorder, Pilates will improve psychic aspects and their physical condition. For all these reasons, the affectation of psychological symptoms will decrease and the quality of life will improve.

ELIGIBILITY:
Inclusion Criteria:

* 1) clinical diagnosis of EDs in the aforementioned hospital;
* 2) aged from 10 to 17 years old;
* 3) written informed consent by the patients and their legal guardians

Exclusion Criteria:

* 1) have other diagnoses of mental illness or
* 2) consumption of narcotic toxins

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Changes in psychopathology - Eating Disorder Inventory-3 (EDI-3). | 3 times (week 0, week 10, week 20).
  EDI-3 (Garner, 2004) is a self-report questionnaire that assesses the presence of eating disorders. The EDI-3 is composed of 91 items, organized into 12 main scales: 3 specific scales of eating behavior disorders (Drive for Thinness, DT; Bulimia, B; Body Dissatisfaction, BD) and 9 general psychological scales that are highly relevant, but not specific to eating disorders (Low Self-Esteem, LSE; Personal Alienation, PA; Interpersonal Insecurity, II; Interpersonal Alienation, IA; Interoceptive Deficits, ID; Emotional Dysregulation, ED; Perfectionism, P; Asceticism, A; Maturity Fears, MF). It also provides 6 composite scores: a specific one of the ED and 5 indices of integrative psychological constructs. The format of six-point Likert-scale responses: always, usually, often, sometimes, rarely or never. The score is between 0 and 4 points. The higher the score, the greater the disorder.
Changes in energy expenditure - SenseWear Mini (SWM). | 3 times (week 0, week 10, week 20).
  SenseWear Mini is a multi-sensor activity monitor that combines tri-axial accelerometry with physiological measurements (skin temperature, heat flux and galvanic skin response) for the estimation of several activity parameters. The information of the different sensors, together with the personal characteristics of the participant (sex, age, height, body weight and the use of hands) is processed through proprietary algorithms of the SenseWear software to estimate the energy expenditure, intensity of physical activity and the number of steps on a minute-by-minute basis.
Changes in body composition - InBody 770 (Body Composition Analyzer). | 3 times (week 0, week 10, week 20).
  InBody 770 (Inbody Co., LTD, Seoul, Korea) to measure body composition through bioelectrical impedance analysis (BIA). Parameters evaluated: Weight (kg); Total Body Water (L); Protein (kg); Minerals (kg); Body Fat Mass (kg); Soft Lean Mass (kg); Fat Free Mass (kg); Skeletal Muscle Mass (kg); Body Mass Index (kg/m2); Percent Body Fat (%); Bone Mineral Contect (kg).
Changes in physical fitness - ALPHA-Fitness Battery. | 3 times (week 0, week 10, week 20).
  ALPHA-Fitness Battery (Assessing Levels of Physical Activity and Fitness) was developed to provide a set of valid, reliable, safe and feasible field tests, in order to assess the physical fitness related to health in children and adolescents, and thus be used in a consensual manner in the Public Health system of the different member states of the European Union. There are three versions of the ALPHA-Fitness battery slightly different depending on the time available for the administration of the tests. We used the extended ALPHA-Fitness Battery. This version of the battery includes handgrip strength, standing broad jump, 4x10 m shuttle run test and 20 m shuttle run test (Ruiz et al., 2011).
Changes in body perception - The Contour Drawing Rating Scale (CDRS). | 3 times (week 0, week 10, week 20).
  The Contour Drawing Rating Scale (CDRS) (Thompson & Gray, 1995) is a scale that evaluates the alterations of the body image. This instrument is a graphic scale, self-administered application, composed of nine female figures views from the front. The person is asked to indicate which figure represents their current body image (perceived body image) and what figure they would like to have (desired body image). The discrepancy between these two classifications represents a measure of body dissatisfaction. The degree of discrepancy varied between -8 and -1 for those who desire a thinner form and between 1 and 8 for those who desire a larger form. A score of 0 was interpreted as satisfaction with body image (Dion et al., 2015). On the other hand, the body image perception index is determined by the following formula: (Estimated size / Actual size) x 100, which would indicate over-estimation when the scores are greater than 100 and underestimation when they are less than 100.
Changes in the quality of life - KIDSCREEN-27. | 3 times (week 0, week 10, week 20).
  KIDSCREEN-27 is a self-administered questionnaire that assesses the health and subjective well-being of children and adolescents (between the ages of 8 and 18) (Ravens-Sieberer et al., 2007). This questionnaire is composed of five dimensions on the Rasch scale: physical well-being, psychological well-being, autonomy and parent relation, peers and social support and school environment. The responses were evaluated and analyzed according to standard algorithms. The recommended syntax steps were performed, including the transformation of Rasch person parameter estimates into Z values, obtaining scale scores as T values with mean scores (± SD) of 50 ± 10 that define normality for children and adolescents of 8-18 years in Europe. Higher scores indicate a higher HRQoL.
Changes in perceived physical fitness - The International Fitness Scale (IFIS). | 3 times (week 0, week 10, week 20).
  The International FItness Scale (IFIS) is a questionnaire that evaluates the physical fitness, of self-administered application, quickly and easily (Ortega et al., 2011). It consists of 5 items (general physical fitness, cardiorespiratory fitness, muscular strength, speed/agility and flexibility) and each with 5 possible Likert-scale responses: "very poor", "poor", "average", "good" or " very good".
Changes in sleep quality - Pittsburgh Sleep Quality Index for adolescents and young adults in Spanish version (AYA-PSQI-S | 3 times (week 0, week 10, week 20).
  Pittsburgh Sleep Quality Index for adolescents and young adults in Spanish version (AYA-PSQI-S) (de la Vega et al., 2015) is a questionnaire slightly adapted from the original (Buysse, Reynolds C. F., Monk, Berman, & Kupfer, 1989) to evaluate the subjective perception of sleep quality in the adolescent population. It consists of 19 items that are grouped into 7 dimensions: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The score of each component ranges from 0 (no difficulty) to 3 (severe difficulty) and the sum of all gives a total score that ranges from 0-21. A high score indicates poor sleep quality and less than 5 is considered high quality.

SECONDARY OUTCOMES:
Changes in blood parameters measured in mg/dL. | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in mg/dL were analyzed: glucose; total cholesterol; triglycerides; prealbumins; transferrin; urea; creatinine; calcium; phosphorus; magnesium; potassium; creatinine kinase; testosterone.
Changes in blood parameters measured in g/dL. | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in g/dL were analyzed: total proteins; albumins; hemoglobin; mean corpuscular hemoglobin concentration.
Changes in blood parameters measured in 10^3/μL. | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in 10^3/μL were analyzed: platelets; red blood cells; leukocytes; lymphocytes; neutrophils; monocytes; basophils; eosinophils.
Changes in blood parameters measured in % | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in % were analyzed: hematocrit; red blood cell dispersion; transferrin saturation index.
Changes in blood parameters measured in fL. | 3 times (week 0, week 10, week 20).
  The following blood parameter measured in fL were analyzed: mean corpuscular volume.
Changes in blood parameters measured in μg/dL | 3 times (week 0, week 10, week 20).
  The following blood parameter measured in μg/dL were analyzed: iron.
Changes in blood parameters measured in mmol/L. | 3 times (week 0, week 10, week 20).
  The following blood parameter measured in mmol/L were analyzed: sodium.
Changes in blood parameters measured in ng/dL | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in ng/dL were analyzed: ferritin; vitamin D; thyroxine; prolactin.
Changes in blood parameters measured in μUI/mL. | 3 times (week 0, week 10, week 20).
  The following blood parameter measured in μUI/mL were analyzed: thyrotropin.
Changes in blood parameters measured in mUI/mL. | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in mUI/mL were analyzed: follitropin; lutropin.
Changes in blood parameters measured in pg/mL. | 3 times (week 0, week 10, week 20).
  The following blood parameters measured in pg/mL were analyzed: estradiol.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garner D. Eating Disorder Inventory-3: Professional manual. Lutz, FL: Psychological Assessment Resources, Inc; 2004.
- [Background] Ruiz JR, Castro-Pinero J, Espana-Romero V, Artero EG, Ortega FB, Cuenca MM, Jimenez-Pavon D, Chillon P, Girela-Rejon MJ, Mora J, Gutierrez A, Suni J, Sjostrom M, Castillo MJ. Field-based fitness assessment in young people: the ALPHA health-related fitness test battery for children and adolescents. Br J Sports Med. 2011 May;45(6):518-24. doi: 10.1136/bjsm.2010.075341. Epub 2010 Oct 19. PMID 20961915
- [Background] Thompson MA, Gray JJ. Development and validation of a new body-image assessment scale. J Pers Assess. 1995 Apr;64(2):258-69. doi: 10.1207/s15327752jpa6402_6. PMID 7722852
- [Background] Dion J, Blackburn ME, Auclair J, Laberge L, Veillette S, Gaudreault M, Vachon P, Perron M, Touchette E. Development and aetiology of body dissatisfaction in adolescent boys and girls. Int J Adolesc Youth. 2015 Apr 3;20(2):151-166. doi: 10.1080/02673843.2014.985320. Epub 2014 Dec 3. PMID 25931646
- [Background] Ravens-Sieberer U, Auquier P, Erhart M, Gosch A, Rajmil L, Bruil J, Power M, Duer W, Cloetta B, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. The KIDSCREEN-27 quality of life measure for children and adolescents: psychometric results from a cross-cultural survey in 13 European countries. Qual Life Res. 2007 Oct;16(8):1347-56. doi: 10.1007/s11136-007-9240-2. Epub 2007 Aug 1. PMID 17668292
- [Background] Ortega FB, Ruiz JR, Espana-Romero V, Vicente-Rodriguez G, Martinez-Gomez D, Manios Y, Beghin L, Molnar D, Widhalm K, Moreno LA, Sjostrom M, Castillo MJ; HELENA study group. The International Fitness Scale (IFIS): usefulness of self-reported fitness in youth. Int J Epidemiol. 2011 Jun;40(3):701-11. doi: 10.1093/ije/dyr039. Epub 2011 Mar 24. PMID 21441238
- [Background] de la Vega R, Tome-Pires C, Sole E, Racine M, Castarlenas E, Jensen MP, Miro J. The Pittsburgh Sleep Quality Index: Validity and factor structure in young people. Psychol Assess. 2015 Dec;27(4):e22-7. doi: 10.1037/pas0000128. PMID 26653055
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771